CLINICAL TRIAL: NCT06761612
Title: A Longitudinal Assessment of Serology and Effectiveness to Determine COVID-19 Vaccine Correlates of Risk (CoR) and Correlates of Protection (CoP) in a Heterogeneous US Population Through Use of Decentralized Sites and Approaches for Data/Specimen Collection
Brief Title: Retail COVID-19 Study
Status: Active, not recruiting | Type: Observational
Sponsor: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: RRPV-24-02-Retail-009
Record Dates: First submitted 2024-12-05; First posted 2025-01-07 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-03

CONDITIONS: COVID - 19
Keywords: Covid-19; Vaccines; Correlates of Protective Immunity; Retail Pharmacy; Walgreens; Observational
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Primary Cohort: Cohort Provides blood draws during on-study visits
  Interventions: Biological: FDA approved mRNA vaccines
- PBMC Cohort: Up to 80 participants providing PBMCs
  Interventions: Biological: FDA approved mRNA vaccines

INTERVENTIONS:
Biological: FDA approved mRNA vaccines — This study is non-interventional as participants will have received an FDA approved mRNA COVID-19 vaccine prior to entering the study. The study protocol does not determine or allocate receipt of vaccine

SUMMARY:
Despite the availability of vaccines, there remains a need to identify specific immune responses that correlate with protection against SARS-CoV-2 infection. Additionally, the operational capability of retail pharmacy infrastructure to collect longitudinal data and biological samples needs to be assessed. This study aims to fill these gaps by determining correlates of protection (CoP), assessing the infrastructure's capability, and examining demographic and geographic differences in participation.

DETAILED DESCRIPTION:
This multi-center study will utilize a prospective, longitudinal observational design to assess CoR and CoP for COVID-19 vaccinations. Prior to enrollment in this study, participants will receive a federally licensed and authorized vaccine, manufactured by Pfizer-BioNTech or Moderna, for the prevention of COVID-19. Each participant will complete a pre-screener questionnaire which will collect information to confirm the participant's eligibility. Upon passing the pre-screener, the participant will complete their electronic consent form and will be enrolled in the study within 72 hours of their vaccination with blood collected to establish baseline for humoral immune marker. A subset of total enrollment, a cohort of 80 participants, will also enroll in the PBMC cohort; participants in the PBMC cohort will enroll in the study within 24 hours of their vaccination with blood collected to establish baseline immune marker levels.

During this study, participants will complete five (5) visits on site (Day 01, Day 31, Day 91, Day 181, Day 366), which will involve data collection and a blood draw. Participants enrolled in the PBMC cohort will have an additional blood draw at Day 01, Day 31, Day 181, and Day 366.

All study participants will complete a weekly electronic patient reported outcome (ePRO) to report symptoms of COVID-19, and to report if they have been exposed to anyone who has tested positive for COVID-19.

Participants will be asked to report to the clinic for a nasal swab test (via molecular assay) when: participant has at least one symptom with or without a fever, and/or if the participant has recent exposure or close contact to another person with COVID-19.

This study aims to enroll at least 90 COVID-19 endpoint cases, based on an annual incidence rate of 2.5%.

ELIGIBILITY:
Inclusion Criteria:

1. People ≥3 years of age at time of enrollment.
2. Willing and able to provide informed consent, or assent in pediatric population, if appropriate, prior to initiation of study procedures.
3. Able to understand and comply with planned study procedures.
4. Available for all study data collection points.
5. Receipt of the most recent FDA-licensed and authorized COVID-19 vaccine (i.e., the 2024-2025 Moderna COVID-19 vaccine or the 2024-2025 Pfizer-BioNTech COVID-19 vaccine which includes the KP.2 strain of the JN.1-lineage vaccine), as recommended by the FDA's Vaccines and Related Biological Products Advisory Committee (VRBPAC) and outlined in the FDA's updated guidance, administered within 3 days of enrollment.

PBMC cohort only:

People ages ≥18 years at time of enrollment. Available for first blood sample collection within 1 day of vaccine.

Exclusion Criteria:

1. Currently participating or plans to participate in another clinical trial involving an investigational product before completing this study.
2. Planned to receive another COVID-19 vaccine within 180 days.
3. Receipt of COVID-19 vaccination within 180 days prior to current vaccination.
4. Receipt of Shingrix vaccine in the 28 days prior to the COVID-19 vaccination or planned receipt of Shingrix vaccine within 28 days after receipt of COVID-19 vaccination.
5. Self-report of recently confirmed COVID-19 infection within 30 days.
6. Any disease or medical condition that, in the opinion of the principal investigator or sub-investigator, is a contraindication to study participation.

PBMC cohort only:

Confirmed positive urine pregnancy test at study visits per Schedule of Activities.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Prior to enrollment in this study, participants will receive a federally licensed and authorized vaccine, manufactured by Pfizer-BioNTech or Moderna, for the prevention of COVID-19. Each participant will complete a pre-screener questionnaire which will collect information to confirm the participant's eligibility. Upon passing the pre-screener, the participant will complete their electronic consent form and will be enrolled in the study within 72 hours of their vaccination with blood collected to establish baseline for humoral immune marker. A subset of total enrollment, a cohort of 80 participants, will also enroll in the PBMC cohort; participants in the PBMC cohort will enroll in the study within 24 hours of their vaccination with blood collected to establish baseline immune marker levels.
Sampling Method: Non-Probability Sample
Enrollment: 2660 (Estimated)
Dates: Start 2024-10-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Serum S protein-specific binding antibody (bAb) concentrations (peak and exposure proximal assessments) Serum SARS-CoV-2 specific neutralizing antibody (nAb) titers (peak and exposure proximal assessments); | Day 1, Day 31, Day 91, Day 181, and Day 366 (i.e., visits 1-5)
  Correlates of Protective Immunity
Valid Viable specimens for SARS-CoV-2 testing | Day 1, Day 31, Day 91, Day 181, and Day 366 (i.e., visits 1-5).
  Number of viable specimens collected at retail pharmacies or retail clinics over the Day 366 follow-up period that meet quality standards required for laboratory analysis.
Number of viable specimens for laboratory analysis | Day 1, Day 31, Day 91, Day 181, and Day 366 (i.e., visits 1-5)
  Viable specimens collected at retail pharmacies or retail clinics that meet quality standards required for laboratory analysis.
Number of valid specimens for CoP testing | Day 1, Day 31, Day 91, Day 181, and Day 366 (i.e., visits 1-5)
  Valid specimens collected at retail pharmacies or retail clinics that meet quality standards required for CoP testing.

SECONDARY OUTCOMES:
Representativeness of number of self-collected nasal swabs and blood specimens | Day 1, Day 31, Day 91, Day 181, and Day 366 (i.e., visits 1-5). Various
  Number of self-collected nasal swabs and blood specimens received over the Day 366 follow-up period overall and stratified by participant demographic and social determinants of health.
Representativeness of Number of valid COVID-19 tests | Day 1, Day 31, Day 91, Day 181, and Day 366 (i.e., visits 1-5)
  COVID-19 resulting in a positive or negative result for SARS-CoV-2 infection overall and stratified by participant demographic and social determinants of health.
Assessment of participant recruitment speed | Day 1, Day 31, Day 91, Day 181, and Day 366 (i.e., visits 1-5)
  Participant recruitment speed measured as time of vaccination to time of enrollment, overall and by site, as well as time to full enrollment overall and stratified by age.
Assessment of participant retention | Day 1, Day 31, Day 91, Day 181, and Day 366 (i.e., visits 1-5)
  Participant retention over study period (from Day 1 through Day 366 follow-up) overall and stratified by age.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Walgreens - 3298 S John Young Pkwy, Kissimmee, Florida
  - Walgreens - 1554 E 55th St, Chicago, Illinois
  - Walgreens - 4385 S Archer Ave, Chicago, Illinois
  - Walgreens - 811 Madison St, Oak Park, Illinois
  - Walgreens - 7251 Lake St, River Forest, Illinois
  - Walgreens - 15100 W 87th Street Pkwy, Lenexa, Kansas
  - Walgreens - 7500 Metcalf Ave, Overland Park, Kansas
  - Walgreens - 215 Beach St, Malden, Massachusetts
  - Walgreens - 17811 E US Highway 24, Independence, Missouri
  - Walgreens - 3845 Broadway Blvd, Kansas City, Missouri
  - Walgreens - 2630 NE Vivion, Kansas City, Missouri
  - Walgreens - 6401 W Charleston Blvd, Las Vegas, Nevada
  - Walgreens - 1445 W Craig Rd, North Las Vegas, Nevada
  - Walgreens - 3218 Atlantic Ave, Atlantic City, New Jersey
  - Walgreens - 520 Convery Blvd, Perth Amboy, New Jersey
  - Walgreens - 420 N Frazier St, Conroe, Texas
  - Walgreens - 1919 W Gray St, Houston, Texas
  - Walgreens - 7440 FM 1960 Rd E, Humble, Texas
  - Walgreens - 8430 Broadway St, Pearland, Texas
  - Walgreens - 3316 Avenue H, Rosenberg, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- See also: Retail COVID-19 Study Website — https://www.retailcovidstudy.com